CLINICAL TRIAL: NCT03324685
Title: A Phase 1 Study to Evaluate the Pharmacokinetic Interaction Potential Between BIIB074 and an Oral Contraceptive Regimen in Healthy Female Subjects
Brief Title: A Drug Interaction Study of BIIB074 and an Oral Contraceptive Regimen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 802HV108
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Drug Interactions
Keywords: Oral Contraceptive, Healthy Volunteers, Ethinyl Estradiol,; Levonorgestrel
MeSH Terms: interventions — vixotrigine; Ethinyl Estradiol; Levonorgestrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BIIB074 150 mg and Oral Contraceptive (Experimental): Participants will receive BIIB074 in tablet form in 150 mg doses every 8 hours on prescription (TID) on days 1-7 and on days 26-32. OC will be taken in tablet form (ethinyl estradiol 30 micrograms and levonorgestrel 150 micrograms) once daily (QD) on days 12-32.
  Interventions: Drug: BIIB074; Drug: OC (ethinyl estradiol and levonorgestrel)

INTERVENTIONS:
Drug: BIIB074 — BIIB074 is administered as specified in the treatment arm.
Drug: OC (ethinyl estradiol and levonorgestrel) — OC is administered as specified in the treatment arm.

SUMMARY:
The primary objective of this study is to evaluate the effect of multiple doses of a uridine diphosphate glucuronosyltransferases (UGT)-inducing oral contraceptive (OC) regimen (ethinyl estradiol and levonorgestrel) on the PK of BIIB074 at steady state; evaluate the effect of multiple doses of BIIB074 on the pharmacokinetics(PK) of an OC regimen (ethinyl estradiol and levonorgestrel) at steady state.

The secondary objective of this study is to evaluate the safety and tolerability of BIIB074 when administered alone and when coadministered with a UGT-inducing OC regimen containing ethinyl estradiol and levonorgestrel and to evaluate the effect of a UGT-inducing OC regimen (ethinyl estradiol and levonorgestrel) on the PK of the M13, M14, and M16 metabolites of BIIB074.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a body mass index between 18 and 32 kg/m^2, inclusive.
* Females of childbearing potential must practice effective non-hormonal contraception during the study and be willing and able to continue contraception for 5 weeks after their last dose of study treatment,
* Must be in good health as determined by the Investigator, based on medical history and screening evaluations.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* History of, or positive test result at Screening for, human immunodeficiency virus (HIV)
* Clinically significant abnormal laboratory test values, as determined by the Investigator, at Screening or Day -1
* Previous intolerance to OC medications
* Other unspecified reasons that, in the opinion of the Investigator or Biogen, make the subject unsuitable for enrollment.

NOTE:Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Hour 0 to Hour 8 (AUC8) for BIIB074 | Day 7, 32
Area Under the Concentration-Time Curve from Hour 0 to Hour 24 (AUC24) for OC | Day 25, 32
Maximum Observed Concentration (Cmax) for BIIB074 | Day 7, 32
Maximum Observed Concentration (Cmax) for OC | Day 25, 32
Time to Reach Maximum Observed Concentration (Tmax) for BIIB074 | Day 7, 32
Terminal Elimination Half-Life (t1/2) of BIIB074 | Day 7, 32
Apparent Clearance (CL/F) for BIIB074 | Day 7, 32
Apparent Volume of Distribution at Steady State (Vss/F) for BIIB074 | Day 7, 32
Time to Maximum Observed Concentration (Tmax) for OC | Day 25, 32
Terminal Elimination Half-Life (t1/2) of OC | Day 25, 32
Apparent Clearance (CL/F) for OC | Day 25, 32
Apparent Volume of Distribution at Steady State (Vss/F) for OC | Day 25, 32

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 71 days
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Number of Participants with Abnormal Change from Baseline in Laboratory Parameters up to Day 33 | Day 3, 7, 24, 28, 33
  Chemistry panel included total protein, albumin, creatinine, blood urea nitrogen, uric acid, bilirubin (total and direct), alkaline phosphatase, ALT, AST, gamma-glutamyl transferase, glucose, calcium, phosphorus, bicarbonate, chloride, sodium, and potassium.
Number of Participants with Abnormal Change from Baseline in Hematology Panel up to Day 33 | Day 3, 7, 24, 28, 33
  Hematology Panel measurements are complete blood count with differential and platelet count, and absolute neutrophil count
Number of Participants with Abnormal Change from Baseline in Urinalysis Panel up to Day 33 | Day 3, 7, 24, 28, 33
  Urinalysis panel included dipstick for occult blood, protein, nitrites, leukocyte esterase, glucose, bilirubin, urobilinogen, ketones, pH, and specific gravity. A microscopic examination will be performed if occult blood, protein, nitrites, or leukocyte esterase is abnormal.
Number of Participants with Abnormal Change from Baseline in Vital Sign Measurements up to Day 33 | Day 1, 3, 7, 12, 24, 25, 26, 28, 33
  Vital signs measurements are temperature, heart rate, systolic and diastolic blood pressure, and respiratory rate
Number of Participants with Abnormal Change from Baseline in Electrocardiogram (ECG) up to Day 33 | Day 1, 3, 7, 12, 25, 26, 28, 33
  12-lead ECGs measurements are heart rate, PR interval, RR interval, QRS duration, QT interval, and QTcF
Number of Participants with Abnormal Change from Baseline in Physical Examination up to Day 33 | Day -1, 33
  Abnormal physical examinations findings that are noted postbaseline and deemed clinically significant by the Investigator will be reported as AEs and will be included in the AE analyses.
AUC 8 of BIIB074 Metabolites M13, M14, and M16 | Day 7, 32
  AUC8 indicates the actual body exposure to BIIB074 metabolites during 8 hours after administration of a BIIB074 dose and is expressed in mg*h/L.
Cmax for BIIB074 Metabolites M13, M14, and M16 | Day 7, 32
  Cmax is the maximum serum concentration that BIIB074 metabolites M13, 14, and 16 achieves in the body after BIIB074 is administered.
Tmax for BIIB074 Metabolites M13, M14, and M16 | Day 7, 32
  Tmax is the amount of time it takes to reach Cmax of the BIIB074 metabolites13,14, and 16 after BIIB074 has been administered.
Terminal Elimination Half-Life (T 1/2) for BIIB074 Metabolites M13, M14, and M16 | Day 7, 32
  The terminal elimination half-life is the time required to divide the plasma concentration of BIIB074 metabolites M13,14,and 16 by two after reaching pseudo-equilibrium.
Metabolite-to-Parent Ratio in AUC (MRauc) for BIIB074 Metabolites M13, M14, and M16 | Day 7, 32
  The MRauc is the ratio of the BIIB074 metabolites M13,14,and 16 to BIIB074 after administration
Number of Participants with Abnormal Change from Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) Assessments | Day 7, 12, 24, 33, and once between Day 39-42
  The C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Daytona Beach, Florida, United States

REFERENCES:
- [Derived] Zhao Y, Versavel M, Tidemann-Miller B, Christmann R, Naik H. Evaluation of the Potential Pharmacokinetic Interactions Between Vixotrigine and an Oral Contraceptive. Clin Drug Investig. 2020 Aug;40(8):737-746. doi: 10.1007/s40261-020-00931-5. PMID 32564301